CLINICAL TRIAL: NCT05701150
Title: AIO-BNHO Comprehensive Clinico-genomics Database Network - AIO-BNHO CONNECT
Acronym: CONNECT
Status: Recruiting | Type: Observational
Sponsor: AIO-Studien-gGmbH (Other)
Collaborators: Daiichi Sankyo Europe, GmbH, a Daiichi Sankyo Company (Industry); Merck Sharp & Dohme LLC (Industry); Janssen-Cilag G.m.b.H (Industry)
Responsible Party: Sponsor
Other Study IDs: AIO-TF-0122
Record Dates: First submitted 2023-01-18; First posted 2023-01-27 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Biospecimen Retention: Samples With DNA — tissue samples collected in clinical routine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MIN Data Set: Patients who did not receive a targeted therapy based on NGS results (outside of a clinical trial)
  Interventions: Other: Minimal documentation; Other: Extended documentation
- EXT Data Set: Patients who received a targeted therapy based on NGS results (outside of a clinical trial)
  Interventions: Other: Extended documentation

INTERVENTIONS:
Other: Minimal documentation — Minimal data documentation only of patients without targeted therapy based on NGS results
  Groups: MIN Data Set
Other: Extended documentation — Extended data documentation of patients with targeted therapy based on NGS results

SUMMARY:
National, retro- and prospective, observational, multicenter clinical research platform to connect clinical and genomic data of patients with advanced (locally advanced, inoperable, or metastatic) solid tumors (excluding NSCLC, SCLC, and mesothelioma) with results from multi-gene next-generation sequencing (NGS) panels (>30 genes)

DETAILED DESCRIPTION:
The AIO-BNHO CONNECT research platform is a clinic-genomic database collecting data on NGS results and corresponding clinical outcomes in patients with advanced solid tumors (excluding NSCLC, SCLC, and mesothelioma). Data of deceased patients will be included. The platform will provide insight into the current state of precision oncology in Germany by compiling real-world data encompassing a broad spectrum of care providers including but not limited to practice-based oncologists, community hospitals, and university hospitals. The platform also comprises a decentral tissue repository with clinically annotated tumor specimens retrieved within routine clinical care that can be used in future collaborative research projects.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of advanced (i.e., locally advanced, inoperable, or metastatic) solid tumor, ineligible for curative surgery and/or curative systemic therapy
* Available results of commercial or non-commercial RNA- and/or DNA-based multi-gene NGS panels with >30 genes analyzed; for non-commercial panels a list of all tested genes and multiple gene biomarkers (e.g., tumor mutational burden (TMB), microsatellite status) must be provided
* Age ≥ 18 years
* Signed and dated informed consent form (not applicable for inclusion of deceased patients)

Exclusion Criteria:

* Diagnosis of NSCLC/SCLC (C34) or mesothelioma (C45)
* NGS results older than two years at the date of patient inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with advanced (locally advanced, inoperable, or metastatic) solid tumors (excluding NSCLC, SCLC, and mesothelioma) ineligible for curative treatment and with results available from multi-gene next-generation sequencing (NGS) panels (>30 genes)
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2022-12-08 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Molecular tumorboard utilization | 3 years
  Proportion of patients who's case was discussed in a Molecular tumorboard
Treatment reality after NGS analysis | 3 years
  Proportion of patients who received at least one targeted therapy based on NGS results, who exclusively received therapies other than targeted therapies based on NGS results or who did not receive any therapy
NGS | 3 years
  Genomic alterations identified by multi-gene NGS panels
Molecular tumorboard | 3 years
  Descriptive analysis of MTB-based therapy recommendations, their implementation rate and reasons for non-implementation
Overall response rate | 3 years
  Overall response rate of targeted therapy based on NGS results
Progression-free survival (PFS) | 3 years
  Progression-free survival from start of targeted therapy based on NGS results
Overall survival | 3 years
  Overall survival from start of targeted therapy based on NGS results
PFS ratio | 3 years
  PFS interval associated with targeted therapy(ies) administered after NGS analysis divided by the time to progression (TTP) interval associated with the last prior treatment(s)

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (3):
  - Praxis für interdisziplinäre Onkologie & Hämatologie, Freiburg im Breisgau, Baden-Wurttemberg
  - Medizinische Fakultät Mannheim der Universität Heidelberg, Mannheim, Baden-Wurttemberg
  - Klinikum der Universität München, München, Bavaria